CLINICAL TRIAL: NCT02501044
Title: Oxygen Desaturation During Hemodialysis: Clinical Correlates and Association With Adverse Outcomes
Brief Title: Oxygen Desaturation During Hemodialysis
Status: Completed | Type: Observational
Sponsor: Renal Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 14-446
Record Dates: First submitted 2015-07-09; First posted 2015-07-17 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Renal Disease; Hypoxia
MeSH Terms: conditions — Kidney Diseases; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Hemodialysis Patients

SUMMARY:
Hemodialysis patients may experience drops in blood oxygen saturation during the hemodialysis treatment, which may lead to hypoxia in the tissues.

The investigators hypothesize that:

1. The cumulative number, severity, or other characteristics of such deoxygenation episodes may be a predictor of adverse outcomes in hemodialysis patients.
2. There may be demographic, anthropometric, clinical, treatment prescription, lab analytical, and other parameters that correlate with the number and severity of deoxygenation episodes and, therefore, may be used for risk stratification. Further, some of these parameters may be modifiable.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patient

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal Research Institute hemodialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 5500 (Actual)
Dates: Start 2012-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Cumulative number of deoxygenation episodes | Up to 36 months
  Crit-Line III monitor recordings (which contain oxygen saturation data) will be extracted from the RRI database and the cumulative number of deoxygenation episodes will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kotanko, MD, Principal Investigator — Renal Research Institute
Locations (1):
- Renal Research Institute, New York, New York, United States